CLINICAL TRIAL: NCT03886116
Title: Effect of Pre-operative Forearm Exercises on Arterial Venous Fistula Maturation and Blood Flow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/2573
Record Dates: First submitted 2019-03-14; First posted 2019-03-22 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: End Stage Renal Disease; Arteriovenous Fistula
Keywords: Arteriovenous Fistula; AVF Maturation; Pre Operative exercise
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): Patient randomized are required to squeeze a soft ball 10 times for a set. They are required to perform 3 sets of 10 squeezes each at a 1 Minute interval.
  3 sets of exercises to be performed twice in the Morning and Evening, for a total of 6 weeks.
  Interventions: Other: Exercise
- No Exercise (No Intervention): Patient is not required to do any exercise.

INTERVENTIONS:
Other: Exercise — 3 sets of 10 forearm exercises performed twice in the Morning and Evening for 6 weeks.
  Arms: Exercise

SUMMARY:
This study will investigate the effect of pre-operative exercise on hemodynamics in the fistula artery and vein, Pre and Post Arteriovenous Fistula Formation as well as the suitability of Cannulation of Arteriovenous Fistula at 12 weeks Post Surgery.

This is a randomised control study with 20 patients each in the Control arm (Group A) or the Exercise arm (Group B). The subjects will be randomised into 1:1 into one of the two groups.

The patients will have an ultrasound doppler vein mapping done prior surgery and the necessary follow up visits.

DETAILED DESCRIPTION:
The incident and prevalent population on renal replacement therapy for End Stage Renal Disease (ESRD) is steadily increasing in Singapore as well as other countries worldwide. Around 85 - 90% of the prevalent dialysis population is on Hemodialysis and Arteriovenous Fistula (AVF).

AVF is considered the Gold standard for safe and effective vascular access for hemodialysis treatment due to its low rates of complication. However, Primary Failure rate of AVFs remain high at around 20 - 25% depending on the site of the surgery, contributed by several factors including the diameter of the artery and the vein used for AVF formation.

If Pre-operative exercise improves the hemodynamics of the AVF and aids the maturation rate in our study, it can be incorporated into clinical guidelines to reduce the primary failure rate of AVF.

Even though, there is sufficient evidence to support the beneficial role of the forearm exercises on fistula blood flow and maturation, there are no studies looking at the effects of Pre-Operative Exercise on AVF maturation. Our Study is aiming to fulfil this gap in knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Age >=21 to <= 90.
* Chronic Kidney Failure patients with Estimated Glomerular Filtration Rate (eGFR) less than 20mls/min.
* Haemodialysis is chosen as their modality of renal replacement therapy.

Exclusion Criteria:

* Potential fistula vein diameter <= 3mm (with application of tornique) on initial vein mapping.
* Known Left ventricular ejection fraction of less than 20% on Echo diagram.
* Previous stroke effecting the AVF arm.
* Calcified brachial or radial arteries and/or duplex evidence of stenosis of >= 50%

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change of Diameter of the vein at 5cm, 10cm & 15cm from wrist joint/elbow joint | Baseline, 1 Week Pre-Op, 6 Weeks Post-Op
  Measure with the use of an Ultrasound Doppler
Diameter of the Artery - Brachial & Radial | Baseline
  Measure with the use of an Ultrasound Doppler
Diameter of the Artery used for AVF | 1 Week Pre-Op
  Measure with the use of an Ultrasound Doppler
Change of Blood Flow Rate in the Artery | Baseline, 1 Week Pre-Op, 6 Weeks Post-Op
  Measure with the use of an Ultrasound Doppler
Diameter of the fistula vein at 5cm, 10cm & 15cm from anastomosis | 6 Weeks Post-Op
  Measure with the use of an Ultrasound Doppler
Diameter of the artery 2cm above anastomosis | 6 Weeks Post-Op
  Measure with the use of an Ultrasound Doppler
Suitability for Cannulation | 6 Weeks Post-Op
  Measure with the use of an Ultrasound Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Tang Tjun Yip, Principal Investigator — Singapore General Hospital; Lee Qing Wei Shaun, Principal Investigator — Singapore General Hospital
Locations (1):
- Tang Tjun Yip, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kong S, Lee KS, Kim J, Jang SH. The effect of two different hand exercises on grip strength, forearm circumference, and vascular maturation in patients who underwent arteriovenous fistula surgery. Ann Rehabil Med. 2014 Oct;38(5):648-57. doi: 10.5535/arm.2014.38.5.648. Epub 2014 Oct 30. PMID 25379494
- [Background] Salimi F, Majd Nassiri G, Moradi M, Keshavarzian A, Farajzadegan Z, Saleki M, Nikpoor A, Ghane M. Assessment of effects of upper extremity exercise with arm tourniquet on maturity of arteriovenous fistula in hemodialysis patients. J Vasc Access. 2013 Jul-Sep;14(3):239-44. doi: 10.5301/jva.5000123. Epub 2013 Jan 3. PMID 23283645
- [Background] Uy AL, Jindal RM, Herndon TW, Yuan CM, Abbott KC, Hurst FP. Impact of isometric handgrip exercises on cephalic vein diameter in non-AVF candidates, a pilot study. J Vasc Access. 2013 Apr-Jun;14(2):157-63. doi: 10.5301/jva.5000116. Epub 2012 Dec 12. PMID 23258587
- [Background] Rus RR, Ponikvar R, Kenda RB, Buturovic-Ponikvar J. Effect of local physical training on the forearm arteries and veins in patients with end-stage renal disease. Blood Purif. 2003;21(6):389-94. doi: 10.1159/000073441. PMID 14586181